CLINICAL TRIAL: NCT00375011
Title: Use of the BreathID to Assess Hepatic Metabolic Reserve and to Predict Hepatic Decompensation in Patients With Cirrhosis in Need of Liver Transplantation
Brief Title: Breath Test to Assess Hepatic Metabolic Reserve and to Predict Hepatic Decompensation in Cirrhotics
Status: Terminated | Type: Observational
Why Stopped: Company restructured and protocol restructured. Resubmitted with IDE approval under new company name-Exalenz
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Virginia Commonwealth University (Other); US Department of Veterans Affairs (U.S. Federal Agency); Hadassah Medical Organization (Other)
Other Study IDs: BID CIRR
Record Dates: First submitted 2006-09-10; First posted 2006-09-12 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Cirrhosis
Keywords: MELD-Model of End Stage Liver Disease score; CTP-Child-Turcotte-Pugh score; MEGX-monoethylglycinexylidide-resultant of metabolism of lidocaine; HCC-Hepatocellular carcinoma; HCV-Hepatitis C virus; NASH-Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The three objectives of this trial are:

1. To demonstrate that a decline in hepatic metabolic function as measured by BreathID will correlate with changes in CTP and MELD scores in patients with cirrhosis.
2. To determine the critical value of hepatic metabolic function as measured by BreathID will predict which patients are at risk to develop complications of cirrhosis.
3. To determine the critical value of hepatic metabolic function as measured by BreathID will predict which patients are at risk for liver related mortality.

The hypothesis is that the BreathID breath test will correlate to CTP and MELD scores, and that thresholds can be established that will help predict risk of complications of cirrhosis and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

1. Mortality in patients with chronic liver disease and cirrhosis:

   Chronic liver disease is the 9th most common cause of death in the United States. Unfortunately, mortality secondary to chronic liver disease, cirrhosis and its complications is expected to increase in the future. This is primarily due to the maturation of the Hepatitis C Virus (HCV) epidemic, a rising rate of hepatocellular carcinoma (HCC)and an increasing prevalence of non-alcoholic steatohepatitis (NASH).

   Mortality in patients with chronic liver disease is typically confined to patients with cirrhosis; and the mortality risk in these patients has long been assessed by the Child-Pugh-Turcotte (CTP) score. More recently, the Model of End-Stage Liver Disease (MELD) has been shown to more accurately predict 30 day survival in patients with cirrhosis. The MELD score is now utilized by the United Network for Organ Sharing (UNOS) to prioritize patients awaiting liver transplantation.

   In general, declining liver function and an increase in the CTP and/or MELD scores are precipitated by the complications of cirrhosis; gastrointestinal bleeding from portal hypertension (variceal and non-variceal), ascites, spontaneous bacterial peritonitis (SBP), hepatic encephalopathy (NE), hepato-renal syndrome (types 1 and 2) and HCC. Patients are considered to have stable cirrhosis when they have intact hepatic function and no prior complications of cirrhosis. Such patients have a CTP score of less than 7; reflective of Childs class A cirrhosis. Approximately 3-5% of patients with stable Child class A cirrhosis will develop worsening in hepatic function and/or complications of cirrhosis and decompensate on a yearly basis. In many patients the development of these complications, the deterioration in global liver function and the rise in MELD is a slow gradual process which allows sufficient time for successful transplantation. In contrast, approximately one-third of patients with cirrhosis develop rapid hepatic decompensation a precipitous rise in MELD and die from complications of cirrhosis before they can either be considered for or receive a liver transplant. This observation explains why pre-transplant mortality for patients on the UNOS waiting list is actually greatest in patients with low MELD, not high MELD scores. It is currently believed that such patients have marginal hepatic metabolic capacity or hepatic reserve which both places them at risk for developing complications of cirrhosis and for rapid deterioration when complications occur.
2. Identifying patients with marginal hepatic reserve at risk for complications and decompensation:

   Tests to assess hepatic metabolic function are conducted by administering either intravenously or orally a compound with high hepatic extraction ratio and/or rapid hepatic metabolism. The rate at which the parent compound is removed from the serum or a metabolic product of the parent compound appears in either the blood, urine, breath or saliva reflects hepatic metabolic function. Some of the compounds which have been successfully utilized for this purpose include choline, caffeine, galactose, aminopyrine, erythromycin, lidocaine and methionine and Methacetin [N-(4-Methoxy-phenyl) acetamide]. Previous studies utilizing a battery of liver function tests have demonstrated that these tests correlate with worsening fibrosis and cirrhosis . The hepatic metabolism of lidocaine to monoethylglycinexylidide (MEGX) has been shown to decline with increasing liver fibrosis and with worsening stages of cirrhosis, improve with successful treatment of the underlying liver disease, and to accurately predict which patients with stable cirrhosis awaiting liver transplantation were at risk to develop future hepatic decompensation. Unfortunately, administering lidocaine to perform this test is associated with parasthesias and could precipitate cardiac arrythmias. Thus, while promising as a potential liver function test the use of lidocaine for this purpose has been largely abandoned.
3. BreathID:

Breath testing with 13C labeled substrates provides a safe, non-invasive means for measuring hepatic metabolism. 13C is a stable, non-radioactive isotope which can by incorporated into a specific location within a test substrate so that it would be released when the compound is metabolized by the liver. 13C-compounds utilized for this purpose are administered orally, rapidly absorbed, metabolized by the liver and 13C is is measured in exhaled breath within 20-30 minutes. Hepatic metabolism of the compound is assessed by measuring the ratio of 13C/12C in exhaled breath. The ability to detect, differentiate and quantify 13C and 12C in exhaled CO2 is has been greatly facilitated by the recent development of the BreathID® collection system and analyzer unit. This portable device continuously senses exhaled breath for 13CO2 in real-time through a nasal cannula worn by the patient. The Breath ID devise utilizing a 13C-urea substrate is currently approved by the Food and Drug Administration to test for the presence of H. Pylori infection. The 13C labeled substrate that has been utilized with the Breath ID device to assess liver function is methacetin. Preliminary data has demonstrated that the metabolism of 13C-methacetin declines with increasing hepatic fibrosis in patients with chronic HCV and parallels the clinical course of patients with acute liver failure prior to and after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis determined by liver histology or clinical findings.
2. Age > 18 years

Exclusion Criteria:

1. Known or suspected HCC
2. Hepato-pulmonary syndrome
3. Hepatorenal syndrome (creatinine > 2.5 mg/dl)
4. Refractory ascites (More than 1 paracentesis within the preceding 3 months of enrollment. A single paracentesis performed for diagnostic purposes is not an exclusion)
5. Hyponatremia
6. Prior TIPS placement
7. Prior episode of variceal hemorrhage
8. MELD score >25
9. Any patient whose expected time to liver transplantation is less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis determined by liver histology or clinical findings
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Shiffman, M.D., Principal Investigator — Virginia Commonwealth University; Douglas M Heuman, M.D., Principal Investigator — Department of Veteran Affairs; Maya Margalit, M.D., Principal Investigator — Hadaassah Medical Organization
Locations (3):
- United States (2):
  - Department of Veteran Affairs, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Hoyert DL, Kung HC, Smith BL. Deaths: preliminary data for 2003. Natl Vital Stat Rep. 2005 Feb 28;53(15):1-48. PMID 15779680
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Said A, Williams J, Holden J, Remington P, Gangnon R, Musat A, Lucey MR. Model for end stage liver disease score predicts mortality across a broad spectrum of liver disease. J Hepatol. 2004 Jun;40(6):897-903. doi: 10.1016/j.jhep.2004.02.010. PMID 15158328
- [Background] Bambha K, Kim WR, Kremers WK, Therneau TM, Kamath PS, Wiesner R, Rosen CB, Thostenson J, Benson JT, Dickson ER. Predicting survival among patients listed for liver transplantation: an assessment of serial MELD measurements. Am J Transplant. 2004 Nov;4(11):1798-804. doi: 10.1111/j.1600-6143.2004.00550.x. PMID 15476479
- [Background] Sanyal AJ, Banas C, Sargeant C, Luketic VA, Sterling RK, Stravitz RT, Shiffman ML, Heuman D, Coterrell A, Fisher RA, Contos MJ, Mills AS. Similarities and differences in outcomes of cirrhosis due to nonalcoholic steatohepatitis and hepatitis C. Hepatology. 2006 Apr;43(4):682-9. doi: 10.1002/hep.21103. PMID 16502396
- [Background] Shiffman ML, Saab S, Feng S, Abecassis MI, Tzakis AG, Goodrich NP, Schaubel DE. Liver and intestine transplantation in the United States, 1995-2004. Am J Transplant. 2006;6(5 Pt 2):1170-87. doi: 10.1111/j.1600-6143.2006.01273.x. PMID 16613594
- [Background] Festi D, Capodicasa S, Vestito A, Mazzella G, Roda E, Vitacolonna E, Petrolati A, Angelico M, Colecchia A. Breath tests with stable isotopes: have they a role in liver transplantation? Eur Rev Med Pharmacol Sci. 2004 Jan-Feb;8(1):55-8. PMID 15209156
- [Background] Braden B, Faust D, Sarrazin U, Zeuzem S, Dietrich CF, Caspary WF, Sarrazin C. 13C-methacetin breath test as liver function test in patients with chronic hepatitis C virus infection. Aliment Pharmacol Ther. 2005 Jan 15;21(2):179-85. doi: 10.1111/j.1365-2036.2005.02317.x. PMID 15679768
- [Background] Festi D, Capodicasa S, Sandri L, Colaiocco-Ferrante L, Staniscia T, Vitacolonna E, Vestito A, Simoni P, Mazzella G, Portincasa P, Roda E, Colecchia A. Measurement of hepatic functional mass by means of 13C-methacetin and 13C-phenylalanine breath tests in chronic liver disease: comparison with Child-Pugh score and serum bile acid levels. World J Gastroenterol. 2005 Jan 7;11(1):142-8. doi: 10.3748/wjg.v11.i1.142. PMID 15609414
- See also: BreathID (device used for study) website — http://www.breathid.com